CLINICAL TRIAL: NCT05668962
Title: Restoration of Radioiodine Uptake with Selpercatinib in RET Fusion-Positive Radioiodine-Refractory Thyroid Cancer: a Phase 2 Study Performed in Collaboration with the International Thyroid Oncology Group (ITOG)
Brief Title: Restor. I-131 Upt. + Selpercatinib in RET F-P RAI-R TC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Lori J. Wirth, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-018
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Thyroid Cancer; Thyroid Carcinoma; Metastatic Thyroid Cancer; Follicular Thyroid Cancer; Unresectable Thyroid Gland Carcinoma; Papillary Thyroid Cancer
Keywords: Thyroid Cancer; Thyroid Carcinoma; Metastatic Thyroid Cancer; Follicular Thyroid Cancer; Unresectable Thyroid Gland Carcinoma; Papillary thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — selpercatinib; Iodine-131; Thyrotropin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SELPERCATINIB + I-131 NaI (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Participants will be treated with Selpercatinib for 4 weeks.
  * In the fourth week of treatment, participants will receive a therapeutic dose of I-131 NaI.
    * Those participants in whom radioiodine uptake has been restored may be offered a second 4-week course of selpercatinib plus I-131 NaI treatment
  Interventions: Drug: Selpercatinib; Drug: Sodium Iodine I-131; Drug: rhTSH

INTERVENTIONS:
Drug: Selpercatinib — Selpercatinib Oral, twice daily during initial treatment period (28 Days). A second course of selpercatinib if the participant is demonstrating clinical benefit to the initial course selpercatinib and deemed clinically appropriate by the treating investigator
  Other Names: Retevmo
Drug: Sodium Iodine I-131 — I-131 NaI, oral, is a standard treatment for all types of follicular-derived thyroid cancers, except anaplastic thyroid cancer
  Other Names: I-131; I-131 NaI
Drug: rhTSH — RhTSH injection, dosage per protocol, timing per protocol during the initial treatment period per standard of care.
  Participants may receive a second course of rhTSH if the participant is demonstrating clinical benefit to the initial course rhTSH and deemed clinically appropriate by the treating investigator.
  Other Names: thyrotropin alfa

SUMMARY:
This research is being done to determine the efficacy of selpercatinib to restore radioactive iodine (I-131 NaI) uptake and allow for I-131 treatment in people with RET fusion-positive radioiodine-refractory thyroid cancer.

This research study involves the study drug selpercatinib in combination with standard of care treatments, I-131 and thyrotropin alfa (rhTSH).

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

* This research study involves the study drug selpercatinib in combination with standard of care treatments, I-131 and thyrotropin alfa (rhTSH). Participants receive study treatment for as long as the disease does not worsen (disease progression) for approximately 1 month for up to two courses of treatment, if participants do not experience any unacceptable side effects, and/or until withdrawal of consent.
* Participants will be followed for 2 years from the date of study registration.
* It is expected that about 30 people will take part in this research study/
* This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

  * The U.S. FDA has approved selpercatinib, I-131 and rhTSH as a treatment option for this disease.
  * The combination therapy is investigational as it has not been approved to treat this disease.
* Selpercatinib, I-131 and rhTSH are standard of care treatment options for thyroid cancer. Selpercatinib is a small molecule designed to block the active RET signaling.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically- or cytologically-confirmed follicular-derived nonanaplastic thyroid cancer that is metastatic and/or unresectable AND harbors a known oncogenic RET gene fusion, performed in a Clinical Laboratory Improvement Amendments (CLIA)-certified or equivalently accredited diagnostic laboratory.
* Tumor tissue or liquid biopsy-based next-generation sequencing (NGS), quantitative polymerase chain reaction (qPCR), and fluorescence in situ hybridization (FISH) for RET gene fusion detection will be permitted.
* Participants ≥ 18 years of age must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

  -- Participants 12 to <18 years of age may enroll with either evaluable (i.e. anatomically visible tumor on cross sectional imaging, but tumors do not need to be >1 cm) or measurable disease per RECIST v1.1.
* Participants should have no single tumor deposit exceeding 4.0 cm in the greatest dimension.
* Participants must have RAI-refractory disease, as defined by:

  * The malignant tissue does not concentrate RAI on a whole body scan following radioiodine administration
  * The tumor tissue has lost the ability to concentrate RAI on a whole body scan following radioiodine administration after previous evidence of uptake at any earlier timepoint,
  * RAI is taken up in some but not all tumor deposits on a whole body scan following radioiodine administration and/or
  * There is progressive disease per RECIST v1.1 despite RAI uptake on a whole body scan following radioiodine administration and/or
  * For patients 12 to <18 years of age, there is persistent anatomically visible tumor on cross sectional imaging following prior therapeutic radioiodine administration
* Participants may have received no more than a total cumulative RAI dose for treatment (not including RAI given for diagnostic purposes only) of 500 mCi (18.5 GBq).
* Participants must have asymptomatic or minimally symptomatic disease, as judged by the treating investigator. For example, patients with bone metastasis associated with mild pain not requiring narcotics for pain control, or patients with lung metastasis associated with mild cough that does not limit the participant's activities, may be considered minimally symptomatic. If confirmation of this criterion is needed, discussion with the protocol chairperson is required prior to enrollment.
* Prior external beam radiotherapy is allowed. For participants with disease limited to a prior radiotherapy field, this must be considered measurable per RECIST v1.1.
* Participants may have had no more than one prior systemic therapy for RAI-refractory thyroid cancer, including lenvatinib, sorafenib, or other MKIs. This also includes chemotherapy and/or targeted therapy administered within a clinical trial, but does not include I-131 NaI or levothyroxine. Prior RET-specific kinase inhibitor therapy, such as selpercatinib and pralsetinib, is not allowed.
* At least 28 days must have passed since any prior radiation or major surgery. At least 28 days must have passed since any prior systemic therapy for thyroid cancer, excluding thyroid hormone replacement.
* Participants must be ≥18 years of age. Patients as young as 12 years of age will be allowed if permitted by local regulatory authorities and institutional review boards.

  -- All patients of 12 to < 18 years of age will be asked to provide assent and the legally designated representative will be asked to provide written consent.
* Participants ≥ 16 years of age must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1. Participants 12 to <16 years of age must have a Lansky Performance Score of ≥ 60.
* Participants must have a life expectancy greater than 12 months.
* Participants must have the ability to swallow medications and have no gastrointestinal abnormality that may alter medication absorption.
* Participants must have adequate organ and marrow function as defined below. Bloodwork must be collected within 7 days prior to Cycle 1 Day 1:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count (ANC) ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥9 g/dL
  * total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) OR <3.0 x institutional ULN for participants with Gilbert syndrome
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN OR ≤5 × institutional ULN if the liver has tumor involvement
  * creatinine ≤ institutional ULN OR creatinine clearance ≥30 mL/min
* Participants must have serum potassium, calcium and magnesium levels within institutional range of normal (may be receiving supplements). Bloodwork must be collected within 7 days prior to Cycle 1 Day 1.
* Known human immunodeficiency virus (HIV)-infected participants on effective anti- retroviral therapy with an undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with treated brain metastases are eligible if the patient is asymptomatic AND follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. For example, participants with nonmelanoma skin cancer, carcinoma in situ of the cervix or malignancy diagnosed ≥2 years previously and not currently receiving anticancer treatment are eligible. Patients receiving adjuvant hormone therapy for breast or prostate cancer with no evidence of disease are eligible.
* Participants with known history or current symptoms of cardiac disease or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Selpercatinib may impair fertility in men and women. The effects of selpercatinib on the developing human fetus are unknown. For this reason and because selpercatinib as well as other therapeutic agents used in this trial may be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 6 months after the last dose of study drug. Unless not allowed by local regulations, WOCBP who are abstinent (if this is complete abstinence, as their preferred and usual lifestyle) or in a same-sex relationship (as part of their preferred and usual lifestyle) must agree to either remain abstinent or stay in a same-sex relationship without sexual relations with males. Periodic abstinence (e.g. calendar, ovulation, symptothermal, postovulation methods), declaration of abstinence just for the duration of the trial, and withdrawal are not acceptable methods of contraception. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men with partners who are WOCBP must agree to use a highly effective contraceptive method during treatment with the study drugs and for 6 months following the last dose of study drug.
* WOCBP must have a negative pregnancy test (serum or urine) within 7 days prior to initiating study treatment, and not be breast-feeding within two months prior to study entry, during treatment, and for ≥1 week after the last dose of study therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy, MKI or radiotherapy within 4 weeks.
* Participants who have had I-131 NaI treatment within 12 months.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Participants who are receiving any other investigational agents.
* Participants with symptomatic CNS metastasis or lesions threatening for spinal cord compression are not eligible.
* Participants with clinically significant active cardiovascular disease or history of Torsades de pointes, history of myocardial infarction within 6 months prior to planned start of study treatment, or prolongation of the corrected QT interval by Fridericia's formula (QTcF) >470 msec on more than one ECG during Screening. Correction of suspected drug-induced QTcF prolongation may be attempted at the investigator's discretion if clinically safe to do so.
* Participants with uncontrolled hypertension at screening, as defined by >160/95 mm Hg.
* Participants with uncontrolled hypertension at screening may be re-screened after appropriate medical therapy for hypertension.
* Participants with an active uncontrolled systemic bacterial, viral, or fungal infection or serious ongoing intercurrent illness, such as hypertension or diabetes, despite optimal treatment, a clinical diagnosis or symptoms of interstitial lung disease, or other serious medical conditions which in the medical judgment of the investigator would prevent the patient from safely participating (screening for chronic conditions is not required).
* Participants with uncontrolled symptomatic hyperthyroidism or hypothyroidism.
* Participants with symptomatic hypercalcemia or hypocalcemia.
* Participants with active hemorrhage or at significant risk for hemorrhage.
* Participants who are taking a concomitant medication that is known to cause QTc prolongation ).
* Participants with clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the drug.
* Participants with other uncontrolled serous intercurrent illness that would interfere with the ability to proceed with study therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 Months
  RECIST v1.1 or Nies criteria in adolescents without RECIST-measurable disease The primary endpoint is best overall response (ORR) (CR and PR) at 6 months. The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).Complete Response (CR) Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed CTCAE v5.0 | up to 2 years
  The safety profile of selpercatinib plus I-131 treatment in this patient population, will be evaluated by assessing by the incidence of treatment-related adverse events per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Rate of restoration of I-131 uptake | Initial Treatment Day 28, Re- Treatment Day 28 up 7 months
  The estimated rate of restoration of I-131 uptake in patients with RAI-refractory RET fusion-positive thyroid cancer treated with selpercatinib will be estimated by determining the rate of positive whole body scans performed after I-131 administration.
thyroglobulin biochemical response rate | Initial Treatment Day 1, Day 21, 3 month follow up, 6 month follow up, Re- Treatment Day 1, follow up, up to 2 years
  The estimated best thyroglobulin biochemical response rates will be determined by comparing serial serum thyroglobulin levels taken every 3 months following treatment to that of the pretreatment baseline level in participants with measurable serum thyroglobulin. Best biochemical response is defined as follows: equals normalization of thyroglobulin level; partial response equals
  ≥50% decrease from baseline thyroglobulin; stable disease equals <50% decrease or increase from baseline; and biochemical progression equals ≥50% increase from baseline (each maintained for at least 4 weeks).
Progression Free Survival | time from registration to the earlier of progression or death due to any cause up to 2 years
  Kaplan-Meier Method
Overall Survival | time from registration to death due to any cause or censored at date last known alive up to 2 years
  Kaplan-Meier Method.
Time to subsequent systemic treatment | 6 Months
  Kaplan-Meier Method Time to subsequent systemic treatment in patients with RET fusion-positive RAIrefractory thyroid cancer will also be estimated.
Overall Response Rate-Adolescent | 6 months
  The structural, biochemical, and overall response rate perl [19] for adolescent patients who enroll without measurable disease will be reported descriptively for adolescents who enroll without RECIST measurable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lori J. Wirth, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation